CLINICAL TRIAL: NCT06057038
Title: A Phase 1 Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of GEN1042 Monotherapy and in Combination With Pembrolizumab ± Chemotherapy in Japanese Subjects With Malignant Solid Tumors
Brief Title: A Safety Trial of GEN1042 in Japanese Subjects With Malignant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1042-03; jRCT2031230438 (Registry Identifier: Japan Registry of Clinical Trials (JRCT))
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Malignant Solid Tumor
MeSH Terms: interventions — pembrolizumab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Monotherapy (non-CNS Malignant Solid Tumors): GEN1042 (Experimental)
  Interventions: Biological: GEN1042
- Combination Therapy Cohort 1 [HNSCC]: GEN1042+Pembro+Chemotherapy (Experimental)
  Interventions: Biological: GEN1042; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil
- Combination Therapy Cohort 2 [HNSCC and NSCLC]: GEN1042+Pembro (Experimental)
  Interventions: Biological: GEN1042; Drug: Pembrolizumab
- Combination Therapy Cohort 3 [HNSCC]: GEN1042+Pembro+Chemotherapy (Experimental)
  Interventions: Biological: GEN1042; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil
- Combination Therapy Cohort 4 [HNSCC and NSCLC]: GEN1042+Pembro (Experimental)
  Interventions: Biological: GEN1042; Drug: Pembrolizumab

INTERVENTIONS:
Biological: GEN1042 — Intravenous
  Other Names: GEN1042 (DuoBody®-CD40x4-1BB)
Drug: Pembrolizumab — Intravenous
  Arms: Combination Therapy Cohort 1 [HNSCC]: GEN1042+Pembro+Chemotherapy; Combination Therapy Cohort 2 [HNSCC and NSCLC]: GEN1042+Pembro; Combination Therapy Cohort 3 [HNSCC]: GEN1042+Pembro+Chemotherapy; Combination Therapy Cohort 4 [HNSCC and NSCLC]: GEN1042+Pembro
Drug: Cisplatin — Intravenous
  Arms: Combination Therapy Cohort 1 [HNSCC]: GEN1042+Pembro+Chemotherapy; Combination Therapy Cohort 3 [HNSCC]: GEN1042+Pembro+Chemotherapy
Drug: Carboplatin — Intravenous
  Arms: Combination Therapy Cohort 1 [HNSCC]: GEN1042+Pembro+Chemotherapy; Combination Therapy Cohort 3 [HNSCC]: GEN1042+Pembro+Chemotherapy
Drug: 5-Fluorouracil — Intravenous
  Arms: Combination Therapy Cohort 1 [HNSCC]: GEN1042+Pembro+Chemotherapy; Combination Therapy Cohort 3 [HNSCC]: GEN1042+Pembro+Chemotherapy

SUMMARY:
This study evaluating GEN1042 will include multiple parts. In this study, GEN1042 alone (phase 1a) or GEN1042 in combination with other anticancer drug(s) (phase 1b) will be evaluated in Japanese participants. The main purpose is to assess the safety and tolerability of GEN1042 monotherapy or GEN1042 in combination in Japanese study participants with cancer.

DETAILED DESCRIPTION:
This is an open-label, trial to evaluate the safety and tolerability, pharmacokinetics (PK), pharmacodynamics, and antitumor activity of GEN1042 in Japanese participants with malignant solid tumors. The trial consists of 2 parts: a GEN1042 Monotherapy Dose Escalation Part (phase 1a); and a Combination Therapy Part (phase 1b).

The purpose of Dose Escalation Part (phase 1a) is to evaluate GEN1042 as monotherapy in participants with non-central nervous system (non-CNS) malignant solid tumors.

The Combination Therapy Part (phase 1b) will evaluate GEN1042 in combination with pembrolizumab (pembro) or pembro along with the standard of care (SOC) chemotherapy in participants with head and neck squamous cell carcinoma (HNSCC) and non-small-cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have measurable disease according to RECIST v1.1.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
3. Acceptable organ and bone marrow function.
4. Participant must have a life expectancy of at least 3 months.

Key Exclusion Criteria:

1. Has clinically significant toxicities from previous anticancer therapies.
2. Has rapidly progressing disease.
3. Has a history of noninfectious pneumonitis/interstitial lung disease.
4. Has a history of liver disease.
5. Has had an allogeneic tissue/solid organ transplant or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of GEN1042.
6. Has any history of intracerebral arteriovenous malformation, cerebral aneurysm, or progressive brain metastases or stroke.
7. Has had major surgery within 4 weeks before Screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | During the first cycle (Cycle length = 21 days)
  Toxicities will be graded for severity according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), version (v) 5.0.
Percentage of Participants with Adverse Events (AEs) | From first dose until the end of the treatment (approximately 3 years)
  An AE is any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.

SECONDARY OUTCOMES:
Maximum (Peak) Plasma Concentration (Cmax) of GEN1042 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 years)
Area Under the Concentration-time Curve (AUC) From Time Zero to Last Quantifiable Sample (AUClast) of GEN1042 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 years)
Time to Reach Cmax (Tmax) of GEN1042 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 years)
Number of Participants with Anti-drug Antibodies (ADA) to GEN1042 | up to 3 years
  Serum samples will be screened for ADAs binding to GEN1042 and the titer of confirmed positive samples will be reported.
Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as percentage of participants with a best overall response (BOR) (Complete Response (CR) or Partial Response (PR)) confirmed by a subsequent BOR of CR or PR at least 4 weeks later per response evaluation criteria in solid tumors (RECIST) v1.1 based on investigator assessment.
Duration of Response (DOR) | Up to 3 years
  DOR only applies to participants whose confirmed BOR is CR or PR and is defined as time from the first documentation of objective tumor response (CR or PR) to the date of first disease progression (PD) or death per RECIST criteria v1.1 based on investigator assessment.
Disease Control Rate (DCR) | Up to 3 years
  The DCR is defined as the percentage of participants with BOR of confirmed CR, confirmed PR, or Stable Disease (SD) per RECIST criteria v1.1 based on investigator assessment.
Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the time from Day 1 in Cycle 1 to the first documented progression or death due to any cause per RECIST criteria v1.1 based on investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (3):
- Japan (3):
  - National Cancer Center East, Kashiwa
  - National Cancer Center Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No